CLINICAL TRIAL: NCT06135805
Title: Impact of the Efficacy of Fluocinonide 0.05% Oral Gel in the Treatment of Oral Lichen Planus
Brief Title: Impact of Fluocinonide 0,05% in Oral Lichen Planus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Catania (Other)
Responsible Party: Principal Investigator, Gaetano Isola, Researcher, University of Catania
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 121-30
Record Dates: First submitted 2023-11-13; First posted 2023-11-18 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Oral Lichen Planus
MeSH Terms: conditions — Lichen Planus, Oral

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Comparator: Fluocinonide 0,,05% oral gel (Experimental): Patients were treated with a topical gel of Fluocinonide 0.05%, applied to oral lesions twice daily for 1 month.
  Interventions: Drug: Fluocinonide 0,05% oral gel
- Placebo Comparator: Placebo (Placebo Comparator): Patients were treated with a topical gel of placebo, applied to oral lesions twice daily for 1 month.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fluocinonide 0,05% oral gel — Application of Fluocinonide oral gel on oral syntomatic lesions
  Arms: Active Comparator: Fluocinonide 0,,05% oral gel
Drug: Placebo — Application of placebo oral gel on oral lesions
  Arms: Placebo Comparator: Placebo

SUMMARY:
A double-blind placebo-controlled trial is conducted in order to evaluate the efficacy of Fluocinonide 0,05% and determinate the statistical significance of the outcome variables. Oral cavity lichen is a chronic inflammatory condition affecting the mucosa of the oral cavity , which significantly reduces the quality of life of affected individuals.

DETAILED DESCRIPTION:
A double-blind placebo-controlled study was conducted to evaluate the clinical efficacy of Fluocinonide 0.05% oral gel and determine the statistical significance of outcome variables.

20 patients with Oral Lichen Planus were divided by a randomization system, into two groups: case group treated with Fluocinonide 0.05% oral gel and applied to oral lesions 2 times a day for 1 month and a placebo group as a control group; with 2 months of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Clinical and histologic diagnosis of Lichen Planus Orale;
* Presence of symptoms related to Lichen Planus Orale;
* Clinical follow-up period of at least 12 weeks;
* Acceptance of informed consent

Exclusion Criteria:

* State of pregnancy or lactation; h
* Histologic signs of dysplasia;
* Medications that induce a lichenoid response (ACE inhibitors, β-blockers, etc.);
* Presence of amalgam fillings in the vicinity of lesions;
* Treatment of oral lichen in the previous 6 months from the start of the program;
* Presence of extraoral lesions (genital, skin, etc.);
* Diabetes being treated with oral hypoglycemic drugs;
* History of previous immunodeficiency;
* HIV seropositivity;
* Previous allogeneic bone marrow transplantation;
* Diagnosis of LES or other autoimmune disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2023-08-20 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Assessment of sings | 3 months
  Assessment of sings using the Thongprasom scoring system at baseline and after 2 months

SECONDARY OUTCOMES:
Assessment of symptoms | 3 months
  Assessment of symptoms using the VAS scale at baseline and after 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Gaetano Isola, Principal Investigator — University of Catania
Locations (1):
- AOU Policlinico G. Rodolico, Catania, Italy

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: 3 months
Access Criteria: Pubmed